CLINICAL TRIAL: NCT05253911
Title: Tucatinib in Patients With Locally Advanced or Metastatic HER2-positive Breast Cancer Who Received at Least Two Prior Anti-HER2 Treatment Regimens: a Multicenter, International, Prospective, Non-interventional Study in Germany and Austria (TRACE)
Brief Title: Tucatinib in Patients With Locally Advanced or Metastatic HER2-positive Breast Cancer Who Received at Least Two Prior Anti-HER2 Treatment Regimens.
Acronym: TRACE
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Collaborators: Seagen Germany GmbH (a Pfizer company) (Unknown)
Responsible Party: Sponsor
Other Study IDs: IOM-120465
Record Dates: First submitted 2022-02-01; First posted 2022-02-24 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: HER2-positive Breast Cancer
Keywords: HER2-positive breast cancer; Tucatinib
MeSH Terms: interventions — tucatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All patients will be asked to give additional informed consent agreeing that their routinely collected tumor samples could be used for further translational research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort 1: Patients receiving tucatinib/trastuzumab/capecitabine (=study treatment) in 1st or 2nd palliative therapy line.
  Interventions: Drug: TUKYSA®
- Cohort 2: Patients receiving tucatinib/trastuzumab/capecitabine (=study treatment) in 3rd or 4th palliative therapy line.
  Interventions: Drug: TUKYSA®

INTERVENTIONS:
Drug: TUKYSA® — tucatinib/trastuzumab/capecitabine according to TUKYSA® SmPC.

SUMMARY:
The objective of this non-interventional study (NIS) is to evaluate tucatinib (TUKYSA®) combined with trastuzumab and capecitabine in adult patients with locally advanced or metastatic HER2-positive breast cancer who have been previously treated with at least two anti-HER2 treatment regimens in a real-world setting,

DETAILED DESCRIPTION:
TRACE will collect real-world data on the treatment of tucatinib/trastuzumab/capecitabine in a broad patient population including older patients and patients with more comorbidities as compared to the pivotal trial HER2CLIMB. In contrast to HER2CLIMB, TRACE will also include patients receiving tucatinib/trastuzumab/capecitabine during 1st and 2nd palliative therapy line who were primarily diagnosed with early breast cancer and therefore already have received two prior anti-HER2 based treatment regimens before enrollment. Until today, no reliable data is available for these patient population. TRACE will primarily focus on HRQoL using the validated EORTC QLQ C30 + QLQ-BR23 + EQ-5D-5L questionnaires. Further aims are to evaluate effectiveness and safety in distinct subgroups focusing on effectiveness of tucatinib/trastuzumab/capecitabine in patients who have experienced prior therapies with trastuzumab and neratinib or capecitabine and HER2-targeted TKIs in the neoadjuvant, adjuvant or palliative setting, respectively.

Study sites may retrospectively include patients within 9 weeks (corresponds to 3 cycles) after start of study treatment up to 6 months after activation of respective site. Retrospectively included patients may have already completed study treatment or may have already deceased at the time of inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* Histologically confirmed HER2+ breast cancer with HER2 positivity defined as a 3+ score by immunohistochemistry (IHC) or a positive result by in situ hybridization (ISH), optionally combined with a IHC2+ score.
* Diagnosis of locally advanced or metastatic HER2+ breast cancer, including patients with brain metastases.
* Prior treatment with at least two prior anti-HER2-based regimens.
* Decision for treatment with tucatinib in combination with trastuzumab and capecitabine according to current SmPC of tucatinib either in

  1st/2nd palliative treatment line (Cohort 1) or 3rd/4th palliative treatment line (Cohort 2).
* Progression after or intolerance of last systemic anti-HER2-based therapy.
* Indication for treatment with tucatinib as assessed by the treating physician.
* Signed written informed consent (only if patient is alive at time of inclusion, not applicable for retrospective inclusion of deceased patients).
* Knowledge of German language.
* Other criteria according to current SmPC of tucatinib

Exclusion Criteria:

* Contraindications according to SmPC of tucatinib
* Participation in an interventional clinical trial within 30 days prior to enrolment or simultaneous participation in an interventional clinical trial.
* Treatment with tucatinib/trastuzumab/capecitabine (=study treatment) in 5th or higher palliative therapy line.
* Onset of tucatinib treatment later than 22 days after start of therapy line (in case tucatinib administration is started later than trastuzumab and/or capecitabine for any reason)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with locally advanced or metastatic HER2-positive breast cancer, including patients with brain metastases, who have been previously treated with at least two prior anti-HER2 treatment regimens and with decision for treatment with tucatinib (TUKYSA®) in combination with trastuzumab and capecitabine.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2022-05-21 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Time to deterioration of EORTC global health scale by at least 10 points | Baseline, up to 24 months
  Only for prospectively enrolled patients: Time to deterioration of EORTC global health scale is defined as the time interval between fill-in date of baseline questionnaire and the first decrease in global health scale score ≥ 10-point (compared to baseline). If there was no such decrease, death will serve as event for this analysis, if occurring within 4 months after last filled-in questionnaire.
Changes in the global health scale | Baseline, up to 24 months
  Only for prospectively enrolled patients: Changes in global health is provided by descriptive statistics of the EQ-5D-5L index value, the EQ-5D-5L visual analogue scale, the EORTC QLQ-C30 global health scale and all functional and symptom scores of the EORTC questionnaires.

SECONDARY OUTCOMES:
Time to next systemic treatment (TTNT) | Baseline, up to 5 years
  TTNT (time to next systemic treatment) is defined as time from first administration of any study treatment (i.e., tucatinib/trastuzumab/capecitabine treatment) to start of a subsequent systemic antineoplastic therapy or death, whichever comes first.
Time to local intracranial treatment (TLT) | Baseline, up to 5 years
  TLT (time to local intracranial treatment) is defined as time from first administration of any study treatment to start of a local intracranial therapy, end of a treatment interruption due to isolated intracranial progression, change of treatment strategy or death, whichever comes first. It will be analyzed for patients with isolated intracranial progression after start of study treatment.
Overall response rate (ORR) | Baseline, up to 5 years
  ORR is defined as proportion of patients with any response (partial or complete remission) overall.
Duration of response (DOR) | Baseline, up to 5 years
  DOR is defined as time from first occurrence of any response (complete or partial remission) to progression or death, whichever comes first. Analysis will be conducted in the subset of patients with any response.
Clinical benefit rate (CBR) | Baseline, up to 5 years
  CBR is defined as proportion of patients with complete or partial remission for best response or with stable disease lasting for at least 24 weeks.
Adverse events (AEs) and serious adverse events (SAEs) according to NCI CTCAE | Baseline, up to 30 days after end of tucatinib treatment
  Adverse events (AEs) and serious adverse events (SAEs) as characterized by type, frequency, severity and seriousness
Safety laboratory value: Aspartate aminotransferase (AST) | Baseline, up to 30 days after end of tucatinib treatment
  During tucatinib administration, safety laboratory will be performed according to routine clinical practice. Laboratory values of AST (Aspartate aminotransferase) measured will be documented continuously during tucatinib treatment. Baseline levels of AST will be presented using descriptive statistics.
Safety laboratory value: Alanine aminotransferase (ALT) | Baseline, up to 30 days after end of tucatinib treatment
  During tucatinib administration, safety laboratory will be performed according to routine clinical practice. Laboratory values of ALT (Alanine aminotransferase) measured will be documented continuously during tucatinib treatment. Baseline levels of ALT will be presented using descriptive statistics.
Safety laboratory value: bilirubin | Baseline, up to 30 days after end of tucatinib treatment
  During tucatinib administration, safety laboratory will be performed according to routine clinical practice. Laboratory values of bilirubin measured will be documented continuously during tucatinib treatment. Baseline levels of bilirubin will be presented using descriptive statistics.
Therapy decision making | Baseline
  Frequencies and percentages of parameters affecting therapy choice.
Previous antineoplastic Therapies | Baseline
  Frequency/type of previous systemic antineoplastic treatments (neoadjuvant/adjuvant/palliative)
Previous anti-HER2 regimens | Baseline
  Frequency and type of previous anti-HER2 based regimens
Subsequent antineoplastic therapies | End of treatment, up to 5 years
  Frequency and type of subsequent systemic antineoplastic therapies
Local antineoplastic therapies | Baseline, up to 5 years
  Frequency and type of local antineoplastic therapies (surgeries, radiotherapies) incl. local intracranial therapies
Details on line of treatment for both cohorts | Baseline
  Cohort 1: frequencies and percentages for line of treatment (1st-line or 2nd-line tucatinib treatment) Cohort 2: frequencies and percentages for line of treatment (3rd-line or 4th-line tucatinib treatment)
Treatment Duration | Baseline, up to 5 years
  Treatment duration of study treatment in total and per substance
Dose intensity | Baseline, up to 5 years
  Dose intensity (absolute and relative) for each substance as prescribed by the treating physician
Dose modifications | Baseline, up to 5 years
  Frequency, type and reasons of dose modifications (dose reductions, skipped administrations/delays/interruption) compared to SmPC of tucatinib for each substance.
Therapy management (use of relevant supportive medications) | Baseline, up to 5 years
  Frequency of usage of antidiarrheal drugs for prophylaxis and treatment of tucatinib-induced diarrhea

CONTACTS AND LOCATIONS:
Overall Officials: Anja Welt, PD Dr., Study Chair — Universitätsklinikum Essen, Innere Klinik (Tumorforschung); Rupert Bartsch, Assoc. Prof. PD Dr., Study Chair — Medical University of Vienna
Locations (2):
- Medizinische Universität Wien, Innere Medizin I, Hämatologie und Onkologie, Vienna, Austria
- Universitätsklinikum Essen, Innere Klinik (Tumorforschung), Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No